CLINICAL TRIAL: NCT01466712
Title: Randomized Double-blind Placebo-controlled Crossover Study to Evaluate the Effects of Formoterol and Beclomethasone Dipropionate Combination Therapy on Small Airways Function in COPD Patients.
Brief Title: Evaluate the Effects of Formoterol and Beclomethasone Dipropionate Combination Therapy on Small Airways Function
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: KU Leuven (Other)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Principal Investigator, Marc Decramer, Principal Investigator, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: S53020
Record Dates: First submitted 2011-11-04; First posted 2011-11-08 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: COPD; Emphysema; Small Airway Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema | interventions — Tiotropium Bromide; Formoterol Fumarate; Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tiotropium+formoterol/beclomethasone (Experimental): run-in of 4 weeks with thiotropium cross-over after first treatment period of 4 weeks
  Interventions: Drug: Tiotropium + formoterol/beclometasone
- tiotropium+placebo (Sham Comparator): cross-over cfr arm1
  Interventions: Drug: tiotropium + placebo

INTERVENTIONS:
Drug: Tiotropium + formoterol/beclometasone — Tiotropium 18 µg/dose once daily (handihaler device) + formoterol, fumarate 6µg + beclometasone, dipropionate 100µg / dose (Pressurised inhaler): 2 puffs bid, for one month.
  Other Names: Inuvair (B10356)
  Arms: Tiotropium+formoterol/beclomethasone
Drug: tiotropium + placebo — Tiotropium 18 µg/dose once daily (handihaler device) + placebo (Pressurised inhaler): 2 puffs bid, for one month.
  Other Names: drug code number B10356
  Arms: tiotropium+placebo

SUMMARY:
Inuvair® is a novel fixed combination product used in the treatment of asthma and under clinical development for the treatment of COPD. Thanks to the extrafine particle size, it is able to target the whole bronchial tree, including the small airways and hence, is expected to act in these airways and it may thus be beneficial in COPD in that sense. In COPD, its action on the small airways is not directly demonstrated thus far. By way of contrast, dear evidence is present that treatment with bronchodilators alone does not beneficially alter small airway function. The study hypothesis states that the effects of inhaled corticosteroids or ICS/LABA combinations on small airway is present and can be objectivated.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis COPD according to last updated GOLD guidelines (post- bronchodilator FEV/FVC below 0,70, FEV1 <80% predicted)
* ex-smokers (ie 1 year from the last cigarette) with at least 10 pack years.
* GOLD stage II and III (FEV1 > 30% predicted)
* by preference naïve to inhaled corticosteroids; in those taking inhaled corticosteroids this medication will be stopped 1 month prior to enrollment in the study
* Patients must have proven small airways dysfunction on routine spirometry as reflected by a drop in FEF25-75 and FEF75 of at least 50%. Moreover, patients must have proven small airways dysfunction on MBW as reflected by Sacin >0,120 that is considered abnormal.

Exclusion Criteria:

* Current smoking
* Active COPD exacerbation
* gold stage I and IV

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-11; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Physiologically measured small airway function based on MBW variables (Scond and Sacin) and lung functional variables (N2-washout, studying the plateau of phase III and closing volume). | Before run-in
  After a run-in period of 4 weeks in which all patients will receive Tiotropium 18 pig per day as treatment for their disease, they will be randomized in two groups: one group receiving Tiotropium + placebo and another group receiving Tiotropium + Inuvair 2 puffs bid, for one month. After this treatment period, there will be a wash-out period of 4 weeks (with tiotropium as run-in).
Physiologically measured small airway function based on MBW variables (Scond and Sacin) and lung functional variables (N2-washout, studying the plateau of phase III and closing volume). | at randomization
  After a run-in period of 4 weeks in which all patients will receive Tiotropium 18 pig per day as treatment for their disease, they will be randomized in two groups: one group receiving Tiotropium + placebo and another group receiving Tiotropium + Inuvair 2 puffs bid, for one month. After this treatment period, there will be a wash-out period of 4 weeks (with tiotropium as run-in).
Physiologically measured small airway function based on MBW variables (Scond and Sacin) and lung functional variables (N2-washout, studying the plateau of phase III and closing volume). | at the end of each treatment period of 4 weeks
  After a run-in period of 4 weeks in which all patients will receive Tiotropium 18 pig per day as treatment for their disease, they will be randomized in two groups: one group receiving Tiotropium + placebo and another group receiving Tiotropium + Inuvair 2 puffs bid, for one month. After this treatment period, there will be a wash-out period of 4 weeks (with tiotropium as run-in).

SECONDARY OUTCOMES:
Relate the abnormalities found in tests of small airway function with the findings of probe-based confocal laser endomicroscopy | Before run-in at the end of each treatment period of 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marc Decramer, Md, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Flanders, Belgium